CLINICAL TRIAL: NCT02655900
Title: Use of 3D Ultrasound to Predict Anal Sphincter Defects
Status: Completed | Type: Observational
Sponsor: Croydon University Hospital (Other)
Responsible Party: Principal Investigator, Ranee Thakar, Consultant Obstetrician and Urogynaecologist, Croydon University Hospital
Other Study IDs: 13/LO/0232
Record Dates: First submitted 2015-09-08; First posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Obstetric Anal Sphincter Injury
Keywords: Obstetric anal sphincter injury,; Ultrasound diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Pelvic Floor Ultrasound — Transperineal Ultrasound (3D TPUS) and Endovaginal Ultrasound (3D EVUS)

SUMMARY:
Injury to the muscles of the back passage (anal canal) is a relatively common problem. This injury can result in problems with bowel control later in life and usually occurs during vaginal childbirth (commonly referred to as 3rd and 4th degree perineal tears). Currently women who have sustained injury to the muscles of the back passage undergo an ultrasound scan by inserting a probe 3 to 4 cms into the back passage. This helps to check if the muscle of the back passage has healed i.e is intact or has a defect. The investigators would like to establish whether a 3D ultrasound scan probe placed outside the vagina can identify the defects and hence avoid inserting the probe into the back passage. In addition to getting the above information using 3D ultrasound scan, the investigators would also like to identify injuries to the pelvic floor muscle (levator ani) in these patients. Which can be diagnosed using the 3D ultrasound probe placed outside the vagina (perineum). Women who sustain injury to this muscle are known to develop prolapse later on in life.

ELIGIBILITY:
Inclusion Criteria:

* Women who sustained an obstetric anal sphincter injury referred to the perineal clinic

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women sustained anal sphincter injury during childbirth being followed up ante or postpartum
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic test accuracy of 3D endovaginal (EVUS) and transperineal ultrasound (TPUS) for diagnosing Obstetric Anal Sphincter injurieS (OASIS) | 3 months Postpartum
  To calculate the diagnostic test characteristics (e.g sensitivity, specificity, positive predictive value, negative predictive value and likelihood ratio) to enable comparison of three methods of ultrasound assessment of the anal sphincter following sphincter injury after vaginal delivery

SECONDARY OUTCOMES:
Prevalence of Levator Ani Muscle Injury in women who sustained Obstetric Anal Sphincter Injury | 3 months Postpartum
  To calculate the prevalence of LAM avulsion in women with OASIS

REFERENCES:
- [Derived] Taithongchai A, van Gruting IMA, Volloyhaug I, Arendsen LP, Sultan AH, Thakar R. Comparing the diagnostic accuracy of 3 ultrasound modalities for diagnosing obstetric anal sphincter injuries. Am J Obstet Gynecol. 2019 Aug;221(2):134.e1-134.e9. doi: 10.1016/j.ajog.2019.04.009. Epub 2019 Apr 11. PMID 30981717